CLINICAL TRIAL: NCT01759966
Title: Autonomic Cardiovascular Control After Heart Transplantation
Acronym: AccHeart
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Vegard Bruun Wyller, MD, PhD Dept of Pediatrics, Oslo University Hospital, Norway, Oslo University Hospital
Other Study IDs: 2012/1428
Record Dates: First submitted 2012-12-28; First posted 2013-01-03 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Heart Transplant Recipients
Keywords: Heart transplantation; Autonomic cardiovascular control; Acute rejection; Cardiac allograft vasculopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood samples for analyses of: genomic DNA, RNA-transcription in whole blood, cytokines, cathecholamines, other blood biomarkers
  2. Urine samples for analyses of: catecholamines, cortisol, other urine biomarkers
  3. Saliva samples for analyses of: cortisol
  4. Heart biopsy specimen for analyses of: acute and chronic rejection (routine surveillence procedure)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Heart transplant recipients: Patients receiving orthotopic heart transplant in the enrollment period
- Healthy controls: Healthy control subjects, having the same age and sex distribution as the heart transplant recipients

SUMMARY:
The purpose of this prospective study is to investigate denervation (ie. surgical cutting of autonomic nerves) and re-innervation (ie. growth of autonomic nerves) in heart transplant recipients. More specifically, we focus on:

1. The physiological consequences of denervation, in particular its consequences for clinical symptoms, orthostatic tolerance (ie. the ability to stand upright) and exercise capacity. We hypothesize that denervation has negative consequences for all these factors.
2. The pathological consequences of denervation and reinnervation, in particular its association to acute rejection and coronary artery disease (cardiac allograft vasculopathy, CAV). We hypothesize that reinnervation protects against acute rejection and development of CAV
3. Donor and recipient factors associated with the reinnervation process. We hypothesize that characteristics of the surgical procedure (such as aorta cross-clamp time) as well as the rehabilitation process of the recipient (such as physical activity) impacts on the reinnervation process.

DETAILED DESCRIPTION:
Heart transplantation is annually offered to more than 3500 patients worldwide. In Norway, the number is approximately 30/year, and all transplants are carried out at one single hospital (Oslo University Hospital, Rikshospitalet).

Normally, the heart function is intimately controlled by the autonomic nervous system (ANS), but all nervous connections are lost during the surgical transplantation procedure, and the transplanted heart thus becomes denervated. In time, regrowth of nerves may cause partial reinnervation of the new heart.

Some evidence suggests that reinnervation improves exercise capacity and reduces episodes of acute rejections and the development of cardiac allograft vasculopathy. The purpose of this study is further to investigate the changes over time with respect to all parts of the autonomic nervous system (the sympathetic, parasympathetic and sensoric part), and the associated physiological and pathological consequences.

The study may provide knowledge which ultimately could help us improve health and quality of live for heart transplant recipients.

ELIGIBILITY:
Inclusion Criteria HTRs:

* Completed heart transplantation during the last 7-12 weeks
* Age > 16 years and < 70 years

Exclusion criteria HTRs:

* Peri- or postoperative complications causing permanent dysfunction of the allograft (such as hyperacute rejection episodes, severe myocardial ischemia, etc.)
* Diabetes with HbA1C > 6,5 % and/or manifest diabetic complications
* Renal failure with plasma creatinine > 200 µmol/L
* ECG abnormalities (scattered ectopic beats ad minor conduction problems are allowed)
* Permanently bed-ridden

Inclusion criteria healthy controls:

- Age and gender matching the HTRs

Exclusion criteria healthy controls:

* Another chronic disease (such as diabetes mellitus)
* Permanent use of pharmaceuticals (including hormone drugs)
* Pregnancy

Ages: 17 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study is to enroll 50 Heart Transplant Recipients (HTRs) and 50 healthy control subjects.
  HTRs are consecutively invited to participate. Baseline investigations are carried out 7-12 weeks after transplantation surgery. Follow-up investigations are scheduled to 6 months and 1, 2 and 3 years after transplantation
  Healthy control subjects will be recruited to matcht the distribution of age and gender among HTRs. The will be examined at one time point only; thus, the healthy controls are not subjected to prospective follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Cardiac allograft vasculopathy | 1 year
  Indications of cardiac allograft vasculopathy (CAV), assessed by intravascular ultrasound (IVUS) during coronary catheterization.
Acute rejections | 1 year
  The frequency of acute rejections episodes and time to first rejection (combined time/event outcome), as assessed by analyses of heart biopsy specimens

SECONDARY OUTCOMES:
Cardiac allograft vasculopathy | 3 years
  Cf. above
Acute rejections | 2 and 3 years
  Cf. above
Autonomic cardiovascular responses | 6 months, 1, 2 and 3 years
  Autonomic cardiovascular responses (such as changes in blood pressures, heart rate, cardiac output, total peripheral resistance and heart rate variability) during head-up tilt-test, valsalva maneuver and isometric exercise
Exercise capacity | 1, 2 and 3 years
  Cardio-pulmonary responses to a standardized exercise tolerance test (treadmill), such as maximal oxygen consumption(maxVO2), heart rate increase, blood pressure increase, etc.
Activity recordings | 6 months, 1, 2 and 3 years
  Number of steps/day during 7 consecutive days, assessed by an accelerometer
Hormonal levels | 6 months, 1, 2 and 3 years
  The levels of catecholamines, cortisol and other hormones influenced by autonomic nervous activity in blood, urine and saliva
General immune activity | 6 months, 1, 2 and 3 years
  The blood levels of cytokines and other markers of immune function, as well as whole blood gene expression.
Pain threshold | 6 months, 1, 2 and 3 years
  Assessment of pain sensitivity by means of an algometer. Anatomically well-defined "trigger-points" are subjected to increasing pressure; the patients alert at the point where the pressure is perceived to be painful
Clinical symptoms | 6 months, 1, 2 and 3 years
  Validated questionnaires assessing: symptoms of autonomic dysfunction, quality of life, pain, fatigue, anxiety, depression and sleep problems.
MetaIodoBenzylGuanidin-scan | 1 and 3 years
  The degree of sympathetic cardiac reinnervation as assessed by the scintigraphic method MetaIodoBenzylGuanidin-scan
Echocardiographic indices | 1, 2 and 3 years
  Echocardiographic indices of cardiac function, such as as systolic and diastolic velocities of the ventricular myocardium based on Tissue Doppler Imaging
Ambulant blood pressure recording | 1, 2 and 3 years
  24 hours ambulant blood pressure recordings
Cardiac catheterization | 1, 2 and 3 years
  Routine data from surveillance cardiac catheterization procedures, such as pressure recordings, angiograms and biopsy assessments

CONTACTS AND LOCATIONS:
Overall Officials: Vegard B Wyller, MD,PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Dept. of Cardiology, Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Christensen AH, Nygaard S, Rolid K, Nytroen K, Gullestad L, Fiane A, Thaulow E, Dohlen G, Saul JP, Wyller VBB. Early Signs of Sinoatrial Reinnervation in the Transplanted Heart. Transplantation. 2021 Sep 1;105(9):2086-2096. doi: 10.1097/TP.0000000000003580. PMID 33323767